CLINICAL TRIAL: NCT06378606
Title: Effect of Screen Based Cognitove Therapy on Mild Dementi in Elderly
Brief Title: Effect of Technology on Cognitive Function in Elderly
Acronym: cogntion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan Hesham Ali (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Nourhan Hesham Ali, physiotherapist /Nourhan Hisham Ali, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004907
Record Dates: First submitted 2024-02-25; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Behavioral Therapy; Cognitive Training

STUDY DESIGN:
Intervention Model Description: The aim of study is to find the effects of screen based cognitive therapy on mild dementia in elderly .
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The aim of study is to find the effects of screen based cognitive therapy on mild dementia in elderly .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): (Therapy group) It will include subjects that will receive computer based cognitive therapy sessions training.
  omega 3 supplement .
  Interventions: Behavioral: cognitive therapy
- Group B (Experimental): (Smartphone group) It will include subjects that will receive home program training by using their smartphones cognitive applications .
  omega 3 supplement .
  Interventions: Behavioral: cognitive therapy
- group c (Placebo Comparator): It won't receive interventions. only omega 3 supplement
  Interventions: Behavioral: cognitive therapy

INTERVENTIONS:
Behavioral: cognitive therapy — intervention : group A: recive computer cognitive traing by rehacom system and omega 3 supplement .
  group B: recive smart phone cognitive application and omega 3 supplement . group c recive omega 3 supplement only.
  Other Names: cognitive training

SUMMARY:
Cognitive technology therapies, including interactive video gaming, computer soft wares and mobile technology, have been used to implement cognitive training and rehabilitation programs. Potential advantages to using technology-based interventions include enhanced accessibility and cost-effectiveness, providing a user experience to be good communicator, immersive and comprehensive.

DETAILED DESCRIPTION:
Aging over 60 years is associated with some progressive decline in cognitive domains, such as processing speed and executive function. A significant decline in cognitive function, particularly memory, which is an early symptom of dementia, can lead to mild cognitive impairment (MCI). Currently it is estimated that 50 million are living with dementia worldwide and nearly 10 million new cases occur every year, representing a serious public health problem. As such, the WHO has suggested that preventing cognitive decline and dementia is a global mental health priority. In addition to impacting the patient, dementia also has a significant impact on the family and society in general. Age is the biggest risk factor for the development of dementia, and aging is associated with a decline of cognitive function. Non-pharmacological interventions such as physical exercise and cognitive interventions may offer an alternative to pharmacological intervention in delaying dementia-related functional decline. Over the last decade, the accessibility and use of computers, smartphones and mobile internet has quickly expanded .

Cognitive technology therapies, including interactive video gaming, computer soft wares and mobile technology, have been used to implement cognitive training and rehabilitation programs. Potential advantages to using technology-based interventions include enhanced accessibility and cost-effectiveness, providing a user experience to be good communicator, immersive and comprehensive.

ELIGIBILITY:
Inclusion criteria

1- Age ≥ 65 years. 2- Literate with ≥ 15 years of education. 3- Older adults with mild dementia. 4- Montreal cognitive assessment score 18-26 .( Pinto et al .,2019). 5- Android smartphone user. 6- Well ability to write and read. Exclusion criteria

1. Major Cardiovascular events , such as Stroke or Myocardial infraction in past three months.
2. Alzheimer's disease.
3. Sever cognitive dementia.
4. Sever hearing difficulty or visual disturbance.
5. Brain injury.
6. Limitation in communications.
7. Chronic kidney diseases.
8. Liver diseases.
9. Low or high educated.
10. Uncontrolled diabetic patients.
11. Thyroid disturbance.
12. Mental and psychological instability .

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive functions assessment | 1 year
  Cognitive function :
  It was assessed by rehacom software and Montreal cognitive assessment (MoCA) which are a highly sensitive and specific screening tool for patients with impaired cognitive function. 1- Rehacom software screening: 9 screening modules detect cognitive functions: 4Attention, 2memory, 1logical reasoning and 2 visual field.
  Montreal test is a short in duration (10- 15 min) 30-point screening test that measures a number of cognitive domains such as visuospatial abilities, executive function, short-term memory, attention/concentration, language, abstract thinking, and orientation. . Patients with MoCA scores of less than 26 are considered cognitively impaired Arabic version was used

SECONDARY OUTCOMES:
Quality of life survey | 1 year
  Quality of life : it was assessed by SF-12 health survey quality of life questionnaire.
  The SF-12 is a generic, standardized questionnaire used to meas- ure two components of HRQoL: physical and mental health. . It is a shorter, yet valid alternative to the most widely used health status scale: the Short-Form-36 Health Survey Questionnaire (SF-36). The SF-12 reproduces the physical and mental component summary scores (PCS/MCS) of the SF-36. In addition, as the SF-12 contains fewer questions and takes less time to complete than the SF-36, it is more appropriate for use with older adults with common geriatric diseases, such as dementia .There scores range from zero (lowest HRQoL)-100 (highest)

CONTACTS AND LOCATIONS:
Overall Officials: ahmed mahdi ahmed, Study Director — Cairo University
Locations (1):
- Nour Ali, Cairo, Giza Governorate, Egypt